CLINICAL TRIAL: NCT07378514
Title: Cobas® Lumira Collection of Venous and Capillary Blood Samples for the Research, Optimization and Calibration of New Diagnostic Devices (EVOLVE)
Brief Title: Cobas® Lumira Collection of Venous and Capillary Blood Samples for the Research, Optimization and Calibration of New Diagnostic Devices
Acronym: EVOLVE
Status: Not yet recruiting | Type: Observational
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: RD007454
Record Dates: First submitted 2026-01-14; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Blood Clots; Infection and Inflammatory Reaction; Heart Disease; Kidney Disease; Vitamin K Antagonist; Diabetes; High Cholesterol; Liver Disease
MeSH Terms: conditions — Thrombosis; Infections; Inflammation; Heart Diseases; Kidney Diseases; Diabetes Mellitus; Hypercholesterolemia; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood and/or plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Blood clot: participants presenting with symptoms indicative of thromboembolic events
  Interventions: Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests
- Infection/Inflammation: participants presenting with symptoms indicative of infection or inflammatory disorders
  Interventions: Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests
- Heart disease: participants presenting with symptoms indicative of heart failure or acute coronary syndrome
  Interventions: Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests
- Kidney disease: participants presenting with symptoms indicative of renal disorders
  Interventions: Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests
- Blood thinners: participants with ongoing vitamin K antagonist therapy for at least four weeks
  Interventions: Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests
- Diabetes: participants with suspected pre-Diabetes or diagnosed with Diabetes Mellitus Type 1 or Type 2
  Interventions: Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests
- High cholesterol: participants presenting with symptoms indicative of Hypercholesterolemia
  Interventions: Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests
- Liver disease: participants with symptoms indicative of hepatic disorders
  Interventions: Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests

INTERVENTIONS:
Diagnostic Test: Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests — Blood samples are obtained and pseudonymized, prior to use for the development, optimization and calibration of diagnostic tests

SUMMARY:
This study is a blood sample collection study, collecting venous and capillary blood samples from adult patients in the UK, with a range of health conditions. The purpose of this study is to collect blood samples to help develop, improve, and fine-tune new and existing diagnostic tests for the cobas® lumira instrument. This instrument is a diagnostic medical device with single-use test strips, that allows diagnostic testing right at the patient's side. The aim is to improve doctors' ability to monitor health conditions more quickly and easily.

Approximately 30,000 patients are expected to participate in this study, across multiple UK sites.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Willing to comply with study procedures.
3. The participant must present as one of the following cohorts (primary presenting condition):

   * Cohort A - Embolism Cohort (participants presenting with symptoms indicative of thromboembolic events)
   * Cohort B - Infection or Inflammation Cohort (participants presenting with symptoms indicative of infection or inflammatory disorders)
   * Cohort C - Cardiovascular Cohort (participants presenting with symptoms indicative of heart failure or acute coronary syndrome)
   * Cohort D - Renal Cohort (participants presenting with symptoms indicative of renal disorders)
   * Cohort E - Oral Anticoagulation Cohort (participants with ongoing vitamin K antagonist therapy for at least four weeks)
   * Cohort F - Diabetes Cohort (participants with suspected pre-Diabetes or diagnosed with Diabetes Mellitus Type 1 or Type 2)
   * Cohort G - Lipid Cohort (participants presenting with symptoms indicative for Hypercholesterolemia )
   * Cohort H - Liver Cohort (participants with symptoms indicative of hepatic disorders).

Inclusion Criteria for Cohorts A, B, C, D, E, G, and H:

1. Participants ≥ 18 years of age

Inclusion Criteria for Cohort F (Diabetes Cohort):

1. Participants ≥ 16 years old

Exclusion Criteria:

1. Subjects deemed inappropriate for the study by the Principal Investigator.
2. Participants who have previously been enrolled in the EVOLVE study in the past 60 days.

Exclusion Criteria for Cohort E (Oral Anticoagulation Cohort):

1. Subjects who are currently taking non-vitamin K antagonist oral anticoagulants (NOACs) including but not limited to apixaban, dabigatran etexilate, edoxaban and rivaroxaban.
2. Subjects who have anti-phospholipid antibody syndrome (APS)
3. The participant is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, experimental drug, or experimental device including either treatment or therapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: UK-based adults presenting to a study site and meeting the eligibility criteria. There are no demographic requirements for this study
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-04 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Biomarker concentration | Baseline
  Blood samples will be used to take a quantitative baseline measurement of 1 or more biomarkers associated with the following health conditions:
  * Thromboembolism
  * Infection/Inflammation
  * Cardiovascular disease
  * Kidney disease
  * Vitamin K antagonist therapy
  * Diabetes
  * Hypercholesterolemia
  * Liver disease.
  Measurements are used for research, development and calibration of point-of-care diagnostic tests, and may compare results between different test methods. There is no statistical analysis planned on these measurements.

IPD SHARING:
Plan to Share IPD: No